CLINICAL TRIAL: NCT00311272
Title: Vaccination With Autologous Dendritic Cells Pulsed With Allogenous Melanoma Lysate (MelCancerVac) for Treatment of Patients With Advanced Colorectal Cancer
Brief Title: Dendritic Cell Vaccination in Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2612-1970
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Colorectal Neoplasms
Keywords: dendritic cells; antigens, neoplasm
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

INTERVENTIONS:
Biological: MelCancerVac

SUMMARY:
Dendritic cells loaded with tumor antigens induce cytotoxic T-cells which have been proved capable of killing both melanoma and breast cancer cells. Melanoma and colorectal cancer cells express some common antigens. Hence it is possible to use melanoma lysate to load the dendritic cells with tumor antigens similar to the antigens expressed by the patients' colorectal cancer cells.

The patient receives 10 vaccinations with 14 days between each. The parameters for effect are changes in tumor/metastasis size measured with computed tomography (CT), decrease in serum concentration of carcinoembryonic antigen (CEA), performance status measured by the World Health Organization (WHO) criteria, and Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* Verified cancer of colon or rectum
* No chemo- or radiation therapy in 6 weeks
* Performance status 0, 1, or 2 (WHO criteria)
* Adequate function of the kidneys, liver, lungs, and heart
* Adequate function of the hematopoietic system and the coagulation system
* Negative pregnancy test and adequate birth control for fertile women

Exclusion Criteria:

* Pregnancy
* Uncontrolled infection

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-11; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Fischer, MD, Principal Investigator — University Hospital Gentofte
Locations (1):
- Surgical Department, University Hospital Gentofte, Hellerup, Denmark

REFERENCES:
- [Derived] Burgdorf SK. Dendritic cell vaccination of patients with metastatic colorectal cancer. Dan Med Bull. 2010 Sep;57(9):B4171. PMID 20816019
- [Derived] Burgdorf SK, Claesson MH, Nielsen HJ, Rosenberg J. Changes in cytokine and biomarker blood levels in patients with colorectal cancer during dendritic cell-based vaccination. Acta Oncol. 2009;48(8):1157-64. doi: 10.3109/02841860903099964. PMID 19863224